CLINICAL TRIAL: NCT06415604
Title: Effects of a Home-based Psychoeducation on Subjective Well-being for Older Adults With Frailty in the Community: A Randomised Controlled Trial
Brief Title: Home-based Psychoeducation for Older Adults With Frailty: A Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TAO An (Other)
Responsible Party: Sponsor-Investigator, TAO An, Mr, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023.585.M
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Frailty; Well-Being, Psychological
Keywords: Subjective well-being; frailty; psychoeducation
MeSH Terms: conditions — Frailty; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will receive 60-minute weekly online group-based psychoeducation sessions for 12 weeks.
  Interventions: Other: Psychoeducation
- Control group (Active Comparator): Participants will receive 60-minute weekly online group-based physical health sessions for 12 weeks.
  Interventions: Other: Attention control

INTERVENTIONS:
Other: Psychoeducation — The content of psychoeducation is based on "Five Ways of Well-being" which covers "Be active", "Connect", "Take Notice", "Keep learning" and "Giving".
  Arms: Experimental group
Other: Attention control — The content of the sessions mainly focuses on physical health information, such as healthy eating, physical exercise, prevention of falls, and pain management.
  Arms: Control group

SUMMARY:
This study aims to examine the effectiveness of a 12-week home-based telerehabilitation programme on improving subjective well-being among community-dwelling older people with frailty.

The main question it aims to answer is

- Could home-based psychoeducation significantly enhance subjective well-being in older adults with frailty in the community?

Participants will receive 12 weekly online group-based sessions at their homes. The content for the experimental group and control group is different:

* Intervention group: psychoeducation
* Control group: physical health education Participants will receive three home visits for data collection. Some of participants in experimental group will receive interview for process evaluation.

ELIGIBILITY:
Inclusion Criteria:

(1) Aged 65 or older; (2) Identified as frail by the FRAIL scale (score ≥3); (3) Mentally competent as determined by the Abbreviated Mental Test (AMT ≥6); (4) Able to speak and understand Cantonese; (5) Living at home; (6) Experienced in using a smartphone (e.g., sending messages, watching videos).

Exclusion Criteria:

(1) Have visual or hearing impairments or language barriers that may impact communication or understanding; (2) Unfit for home-based exercise, as indicated by a score of 1 or higher on the 25-item HOME-FAST, a tool for identifying home fall hazards; (3) Currently engaging in exercise for at least 150 minutes per week over the past four weeks; (4) Undergoing active psychiatric or antidepressant treatment or participating in other physical exercise or rehabilitation programs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Subjective well-being | baseline, 12 weeks post-allocation, 24 weeks post-allocation
  The Chinese 5-item World Health Organization Well-Being Index

SECONDARY OUTCOMES:
Frailty level | baseline, 12 weeks post-allocation, 24 weeks post-allocation
  FRAIL scale
Physical functioning | baseline, 12 weeks post-allocation, 24 weeks post-allocation
  The Senior Fitness Test: It covers four dimensions, including muscle endurance, balance, flexibility, and tolerance measured by 30-sec arm-curl test, 30-sec chair-stand test, back-scratch test, chair sit-and-reach test, 8-foot up-and-go test, two-min step test
Activities of daily living | baseline, 12 weeks post-allocation, 24 weeks post-allocation
  Katz Index of Independence in Activities of Daily Living
Instrumental activities of daily living | baseline, 12 weeks post-allocation, 24 weeks post-allocation
  Lawton Instrumental Activities of Daily Living Scale
Depressive symptoms | baseline, 12 weeks post-allocation, 24 weeks post-allocation
  4-item Geriatric Depression scale
Social support | baseline, 12 weeks post-allocation, 24 weeks post-allocation
  10-item Duke Social Support Index
Quality of life | baseline, 12 weeks post-allocation, 24 weeks post-allocation
  EuroQol 5-Dimension 5-Level

CONTACTS AND LOCATIONS:
Locations (1):
- The Nethersole School of Nursing, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No